CLINICAL TRIAL: NCT06942624
Title: Phage Therapy for the Treatment of a Chronic Enterococcus Faecium Periprosthetic Joint Infection
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orthopaedic Innovation Centre (Other)
Collaborators: Cytophage Technologies Inc. (Unknown); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OIC-Phage-2025-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Periprosthetic Joint Infection
MeSH Terms: interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Lytic phage prepared in injection-grade saline-magnesium buffer will be given via two routes:
  * intravenously twice daily, and concomitantly,
  * intra-articularly twice daily, for a total duration of 14 days.
  In addition to phage therapy, the patient will receive standard of care antibiotic therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phage Therapy (Experimental): Lytic phage prepared in injection-grade saline-magnesium buffer will be given via two routes: a) intravenously twice daily, and concomitantly, b) intra-articularly twice daily, for a total duration of 14 days. In addition to phage therapy, the patient will receive standard of care antibiotic therapy.
  Interventions: Biological: Phage Therapy

INTERVENTIONS:
Biological: Phage Therapy — Our phage is an investigational treatment for bacterial infections. Our lytic phage preparation was provided by Cytophage Technologies (CIP-200).

SUMMARY:
This purpose of this clinical trial is to evaluate the safety, tolerability and efficacy of a bacteriophage therapy in a patient with a methicillin-susceptible Enterococcus faecium (E. faecium) prosthetic joint infection (PJI) of the hip. We have exhausted all surgical and medical management of PJI for our patient.

The phage will be administered to the study patient during a 14 days period via intravenous and intra-articular. The patient will be monitored in clinic for up to 1 year.

DETAILED DESCRIPTION:
This is a single-patient study, to assess a treatment option for a case of a recurrent methicillin-susceptible E. faecium infection in a prosthetic hip joint. The patient has repeatedly failed standard of care medical and surgical management.

Given the severity and chronicity of E. faecium infection and burden of infected hardware, the only option to achieve surgical source control would involve an aggressive, high risk surgical approach: a high amputation of the left leg to remove infected hardware and peri-implant bone and tissues. In the absence of any viable adjunctive antimicrobial therapy, this patient is at high risk of mortality and morbidity. It is therefore paramount that we explore alternative treatment modalities for the management of this infection, such as bacteriophage (phage) therapy.

The primary objective of this study is to investigate the preliminary efficacy, safety, and tolerability of systemic (intravenous) and intra-articular administration of a lytic phage (in our patient with chronic E. faecium PJI.

Secondary objectives will be documenting clinical changes pre- and post-therapy, as well as identifying adjunctive changes in biomarkers (C-reactive protein [CRP], erythrocyte sedimentation rate [ESR], and interleukin-6 [IL-6]) correlated with PJI as well as phage titres.

In this study, lytic phage prepared in injection-grade saline will be administered to the patient both intravenously and intraarticularly, twice a day for a duration of 14 days. In addition to phage therapy, the patient will receive standard of care antibiotic therapy.

The patient will remain in clinical follow-up for up to one year.

ELIGIBILITY:
Inclusion Criteria:

This N-of-1 Phage therapy is designed for one patient who meet the following conditions

* Willingness to provide signed and dated informed consent form to participate in the clinical study
* Chronic prosthetic joint infection
* History of multiple surgical and medication managements with no success

Exclusion Criteria:

* below 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety of phage therapy | Day 0 to 1 year from treatment
  Reactions and adverse events to the treatment
Efficacy of phage therapy | 1 Year
  No recurrence of the infection
Tolerability of phage therapy | Day 0 to Day 13 of treatment
  Reactions and adverse events to the intravenous and intra-articular administration

SECONDARY OUTCOMES:
Changes in biomarkers (C-reactive protein) | Day 0 to 1 year from treatment
  Serum C-reactive protein (mg/L) as measured at baseline
Changes in biomarkers (erythrocyte sedimentation rate) | Day 0 to 1 year from treatment
  Serum erythrocyte sedimentation rate (mm/hr) as measured at baseline
Changes in biomarkers (interleukin-6) | Day 0 to 1 year from treatment
  Serum interleukin-6 (pg/mL) as measured at baseline
Changes in biomarkers (phage titres) | Day 0 to Day 13 of treatment
  Phage particles present in a given volume of liquid (PFU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: David Hedden, MD, Principal Investigator — Concordia Hospital
Locations (1):
- Concordia Hospital, Winnipeg, Manitoba, Canada